CLINICAL TRIAL: NCT01333722
Title: A Randomized, Multicenter Study Comparing the Analgesic Efficacy and Safety of Hydrocodone / Acetaminophen Extended Release to Placebo in Subjects With Acute Pain Following Bunionectomy
Brief Title: Acute Pain Study Following Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M12-169
Record Dates: First submitted 2011-04-11; First posted 2011-04-12 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Hydrocodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): placebo, 1 oral tablet every 12 hours
  Interventions: Drug: Placebo
- Hydrocodone/Acetaminophen Extended Release (Experimental): hydrocodone/acetaminophen extended release, 1 oral tablet every 12 hours
  Interventions: Drug: Hydrocodone/Acetaminophen Extended Release

INTERVENTIONS:
Drug: Hydrocodone/Acetaminophen Extended Release
  Other Names: ABT-712
  Arms: Hydrocodone/Acetaminophen Extended Release
Drug: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
The primary purpose of this study was to evaluate analgesic efficacy and safety of hydrocodone/acetaminophen extended release compared to placebo in the treatment of moderate to severe pain following bunionectomy.

DETAILED DESCRIPTION:
The bunionectomy was performed under regional anesthesia and propofol sedation. Perioperative anesthesia was standardized for all participants. Upon completion of surgery, designated study personnel ensured continued eligibility per the selection criteria of the protocol.

After an appropriate period of time following bunionectomy, participants who had a pain intensity score of ≥ 40 mm on a 100 mm visual analog scale (VAS) and moderate or severe pain intensity per the categorical pain intensity scale were eligible for randomization, in equal numbers, into 1 of 2 treatment arms: hydrocodone/acetaminophen extended release or placebo.

ELIGIBILITY:
Inclusion Criteria:

Subjects who were in general good health, experiencing moderate to severe pain following bunionectomy

Exclusion Criteria:

* Subjects who underwent Base wedge osteotomy and / or Long-Z Hart bunionectomy procedures
* Drug allergies to hydrocodone, acetaminophen
* Clinically significant or uncontrolled medical disorders or illness - history of drug or alcohol abuse / addiction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Quintana Diez, MD, Study Director — AbbVie
Locations (3):
- United States (3):
  - Site Reference ID/Investigator# 51464, Pasadena, California
  - Site Reference ID/Investigator# 51602, Austin, Texas
  - Site Reference ID/Investigator# 51344, Salt Lake City, Utah

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydrocodone/Acetaminophen Extended Release: 1 dose of hydrocodone/acetaminophen extended release tablet, administered once every 12 hours (for a total of 4 doses).
- Placebo: 1 dose of placebo tablet, administered once every 12 hours (for a total of 4 doses).
Period: Overall Study
Arm/Group | Hydrocodone/Acetaminophen Extended Release | Placebo
Started | 51 | 49
Completed | 51 | 46
Not Completed | 0 | 3
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrocodone/Acetaminophen Extended Release | Placebo | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (11.79) | 41.6 (13.85) | 40.3 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 44 | 85
  Male | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference (SPID) Using the Pain Intensity Visual Analog Scale (VAS)
Description: Participants assessed pain intensity on a 100 mm visual analogue scale (VAS) with 0 meaning "no pain" and 100 meaning the "worst pain imaginable". The SPID VAS score for 0 to 12 hours following initial study drug dose measured the cumulative pain intensity difference during treatment with higher mean SPID VAS scores indicating greater improvement from Baseline. The SPID score is a measure of the cumulative pain intensity difference during treatment and the area under the curve was estimated using the linear trapezoidal rule.
Time Frame: From time of first study drug administration to 12 hours following first study drug administration
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Hydrocodone/Acetaminophen Extended Release | Placebo
Number analyzed (Participants) | 51 | 49
scores on a scale | 259.0 (37.52) | 39.4 (38.10)

2. Secondary Outcome: TOTPAR (Total Pain Relief)
Description: TOTPAR was the time-interval weighted sum of pain relief. Pain relief was assessed by participants' responses to how their pain relief was compared with the pain they had just before receiving the first dose of study drug: no relief, a little relief, some relief, a lot of relief, or complete relief. Higher mean TOTPAR scores indicate better pain relief. The TOTPAR score is a measure of the cumulative pain intensity difference during treatment and the area under the curve was estimated using the linear trapezoidal rule.
Time Frame: From time of first study drug administration to 12 hours following first study drug administration
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Hydrocodone/Acetaminophen Extended Release | Placebo
Number analyzed (Participants) | 51 | 49
scores on a scale | 15.4 (1.72) | 5.3 (1.74)

3. Secondary Outcome: SPRID (Pain Relief and Pain Intensity Difference)
Description: SPRID was defined as the sum of Pain Relief score (TOTPAR, See Outcome Measure 2 for details*) plus the Pain Intensity Difference (SPID) Categorical score, where participants assessed pain intensity on a Categorical Pain Intensity Scale by answering the following question: "My pain at this time is…" with one of the following responses: no pain or none, mild pain, moderate pain, or severe pain). Higher mean SPRID scores indicated better pain control. The SPRID score is a measure of the cumulative pain intensity difference during treatment and the area under the curve was estimated using the linear trapezoidal rule.
Time Frame: From time of first study drug administration to 12 hours following first study drug administration
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Hydrocodone/Acetaminophen Extended Release | Placebo
Number analyzed (Participants) | 51 | 49
scores on a scale | 23.4 (2.75) | 7.2 (2.78)

4. Secondary Outcome: Time to Perceptible and Meaningful Pain Relief
Description: The median time (minutes) from first perceptible pain relief (onset of pain relief) and time until first meaningful pain relief.
Time Frame: From time of first study drug administration to 12 hours following first study drug administration
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Hydrocodone/Acetaminophen Extended Release | Placebo
Number analyzed (Participants) | 51 | 49
minutes
  Time to Onset of Perceptible Pain Relief | 34.0 [29.0 to 45.0] | 56.0 [31.0 to 184.0]
  Time to Onset of Meaningful Pain Relief | 119.0 [73.0 to 447.0] | NA [NA to NA] — Not available from Kaplan-Meier estimate.

ADVERSE EVENTS:
Time Frame: AEs were recorded from study drug administration until 30 days following discontinuation of study drug (total 32 days); SAEs were recorded from the time informed consent was obtained until 30 days following discontinuation of study drug (total 51 days).
Arm/Group | Hydrocodone/Acetaminophen Extended Release | Placebo
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/49
Other Adverse Events (participants affected / at risk) | 28/51 | 14/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hydrocodone/Acetaminophen Extended Release (N=51) | Placebo (N=49)
NAUSEA (Gastrointestinal disorders) | 17 | 8
VOMITING (Gastrointestinal disorders) | 8 | 3
CELLULITIS (Infections and infestations) | 4 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 0
DIZZINESS (Nervous system disorders) | 7 | 3
HEADACHE (Nervous system disorders) | 6 | 7
SOMNOLENCE (Nervous system disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.